CLINICAL TRIAL: NCT00673049
Title: Randomized, Open Label, Phase 3 Trial Of Erlotinib Alone Or In Combination With CP-751,871 In Patients With Advanced Non Small Cell Lung Cancer Of Non Adenocarcinoma Histology
Brief Title: Trial Of CP-751, 871 And Erlotinib In Refractory Lung Cancer
Acronym: NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021018
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Carcinoma, Large Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Carcinoma, Adenosquamous Cell
Keywords: IGR-1R; Non small cell lung cancer; CP-751; 871; Figitumumab
MeSH Terms: conditions — Carcinoma, Large Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Carcinoma | interventions — figitumumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): The CP 751,871 treatment in combination with erlotinib will be given in three week cycles.
  CP 751,871 (20 mg/kg) + erlotinib (150 mg/day) CP 751,871 will be administered as an IV infusion on study Days 1 and 2 in Cycle 1, and every three weeks (from Day 1) (Cycle) thereafter.
  Interventions: Drug: CP 751,871 (Figitumumab); Drug: Erlotinib
- Arm B (Active Comparator): Erlotinib (one tablet of 150 mg/day PO). Erlotinib will be taken at least one hour before or two hours after the ingestion of food)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: CP 751,871 (Figitumumab) — CP 751,871 (20 mg/kg) will be administered as an IV infusion on study Days 1 and 2 in Cycle 1, and every three weeks (from Day 1) (Cycle) thereafter.
  Arms: Arm A
Drug: Erlotinib — Erlotinib (one tablet of 150 mg/day PO).
  Arms: Arm A
Drug: Erlotinib — Erlotinib (one tablet of 150 mg/day PO). Erlotinib will be taken at least one hour before or two hours after the ingestion of food.
  Arms: Arm B

SUMMARY:
The objective of this study is to test a clinical benefit of the addition of CP 751,871 to erlotinib therapy in patients with advanced NSCLC of non adenocarcinoma histology. The primary endpoint is Overall Survival (OS).

DETAILED DESCRIPTION:
This study was terminated on March 8, 2010 due to an analysis by an independent Data Safety Monitoring Committee (DSMC) indicating that the addition of CP-751,871 [figitumumab] to erlotinib [Tarceva] would be unlikely to meet the primary endpoint of improving overall survival when compared to erlotinib alone.

This Oncology study continues as terminated, however for ethical reasons some patients, noted with resultant benefit, continue receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non small cell lung cancer with a primary histology of squamous cell, large cell or adenosquamous carcinoma. At least 1 measurable lesion, as defined by RECIST.

Exclusion Criteria:

* Primary NSCLC adenocarcinoma and its subtypes or unknown/unspecified histology.
* Prior Erlotinib therapy.
* Prior anti IGF IR based investigational therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (145):
- United States (56):
  - Pfizer Investigational Site, Fort Smith, Arkansas
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Lakeport, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Petaluma, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Thousand Oaks, California
  - Pfizer Investigational Site, Westlake Valley, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lafayette, Colorado
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Lake City, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Alpharetta, Georgia
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Cumming, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Duluth, Georgia
  - Pfizer Investigational Site, Lake Spivey, Georgia
  - Pfizer Investigational Site, Lawrenceville, Georgia
  - Pfizer Investigational Site, Snellville, Georgia
  - Pfizer Investigational Site, Bloomington, Illinois
  - Pfizer Investigational Site, Peoria, Illinois
  - Pfizer Investigational Site, Beech Grove, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Waterloo, Iowa
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, New Albany, Mississippi
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Manchester, New Hampshire
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Lake Success, New York
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Gloucester, Virginia
  - Pfizer Investigational Site, Glouster, Virginia
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Williamsburg, Virginia
  - Pfizer Investigational Site, Wenatchee, Washington
  - Pfizer Investigational Site, Wheeling, West Virginia
  - Pfizer Investigational Site, Cody, Wyoming
- Belgium (2):
  - Pfizer Investigational Site, Brasschaat
  - Pfizer Investigational Site, Mons
- Brazil (5):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Higienópolis, Sao Paulo/ Brazil
  - Pfizer Investigational Site, Santo André, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (3):
  - Pfizer Investigational Site, Sofia, Bulgaria
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Varna
- Canada (2):
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Independencia, Santiago, RM, Chile
- Czechia (4):
  - Pfizer Investigational Site, Kutná Hora
  - Pfizer Investigational Site, Nová Ves pod Pleší
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Tábor
- France (8):
  - Pfizer Investigational Site, Rennes, Cedex 9
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, La Tronche
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Saint Pierre La Réunion Cedex
  - Pfizer Investigational Site, Saint-Priest-en-Jarez
  - Pfizer Investigational Site, Villejuif
- Greece (2):
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Larissa
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Mátraháza
  - Pfizer Investigational Site, Székesfehérvár
- Indonesia (2):
  - Pfizer Investigational Site, Jakarta, DKI Jakarta
  - Pfizer Investigational Site, Surabaya, East Java
- Ireland (2):
  - Pfizer Investigational Site, Cork
  - Pfizer Investigational Site, Dublin
- Italy (8):
  - Pfizer Investigational Site, Avellino
  - Pfizer Investigational Site, Aviano (PN)
  - Pfizer Investigational Site, Cattolica (RN)
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Orbassano (TO)
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Rimini
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, Riga, Latvia
- Poland (7):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Olsztyn
  - Pfizer Investigational Site, Rybnik
  - Pfizer Investigational Site, Wodzislaw Sl.
- Pfizer Investigational Site, Ponce, PR, Puerto Rico
- Romania (3):
  - Pfizer Investigational Site, Cluj-Napoca, Cluj
  - Pfizer Investigational Site, Cluj-Napoca
  - Pfizer Investigational Site, Iași
- Russia (4):
  - Pfizer Investigational Site, Krasnodar
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Sochi
- Serbia (2):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Kamenitz
- Pfizer Investigational Site, Ljubljana, Slovenia
- South Africa (2):
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Cape Town
- South Korea (2):
  - Pfizer Investigational Site, Gyeonggi-do
  - Pfizer Investigational Site, Seoul
- Spain (9):
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Manresa, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Girona, Girona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Seville, Sevilla
- Switzerland (4):
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Ch-4101 Bruderholz
  - Pfizer Investigational Site, Chur
  - Pfizer Investigational Site, Liestal
- Taiwan (3):
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyuan
- Ukraine (5):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Sumy
- United Kingdom (3):
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- [Derived] Scagliotti GV, Bondarenko I, Blackhall F, Barlesi F, Hsia TC, Jassem J, Milanowski J, Popat S, Sanchez-Torres JM, Novello S, Benner RJ, Green S, Molpus K, Soria JC, Shepherd FA. Randomized, phase III trial of figitumumab in combination with erlotinib versus erlotinib alone in patients with nonadenocarcinoma nonsmall-cell lung cancer. Ann Oncol. 2015 Mar;26(3):497-504. doi: 10.1093/annonc/mdu517. Epub 2014 Nov 13. PMID 25395283
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021018&StudyName=Trial%20Of%20CP-751%2C%20871%20And%20Erlotinib%20In%20Refractory%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab + Erlotinib (Randomized to and Treated With): Figitumumab ( [CP-751,871], figi) was given in combination with erlotinib (erlo) in 3-week cycles. Figitumumab 20 milligram/kilogram (mg/kg) was administered as an intravenous (IV) infusion on Days 1 and 2 in Cycle 1, and on Day 1 every 3 weeks (from Day 1) thereafter. Erlotinib was taken as 150 milligram (mg) daily at least 1 hour before or 2 hours after the ingestion of food.
- Erlotinib (Randomized to and Treated With); Randomized to Figi + Erlo Arm But Treated Only With Erlo: Erlotinib was taken as 150 mg daily at least 1 hour before or 2 hours after the ingestion of food.
- Erlotinib, Then Figitumumab: Figitumumab 20 mg/kg was given as a single-agent therapy to participants who had disease progression on erlotinib alone. Figitumumab was administered in 3-week cycles as IV infusion on study Days 1 and 2 in Cycle 1, and on Day 1 every 3 weeks (from Day 1) thereafter.
Period: Before Progression on Erlotinib
Arm/Group | Figitumumab + Erlotinib (Randomized to and Treated With) | Erlotinib (Randomized to and Treated With) | Randomized to Figi + Erlo Arm But Treated Only With Erlo | Erlotinib, Then Figitumumab
Started | 292 | 290 | 1 | 0 (Participants treated with erlo alone who subsequently received figi upon disease progression.)
Treated | 289 | 289 | 1 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 292 | 290 | 1 | 0
Not completed — Randomized but not treated | 3 | 1 | 0 | 0
Not completed — Death | 235 | 167 | 1 | 0
Not completed — Lost to Follow-up | 9 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 26 | 18 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0
Not completed — study terminated by sponsor | 18 | 14 | 0 | 0
Not completed — Switched to figitumumab | 0 | 83 | 0 | 0
Period: After Progression on Erlotinib
Arm/Group | Figitumumab + Erlotinib (Randomized to and Treated With) | Erlotinib (Randomized to and Treated With) | Randomized to Figi + Erlo Arm But Treated Only With Erlo | Erlotinib, Then Figitumumab
Started | 0 | 0 | 0 | 83
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 83
Not completed — Death | 0 | 0 | 0 | 71
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5
Not completed — study terminated by sponsor | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Figitumumab + Erlotinib (as Randomized): Figitumumab (20 mg/kg) in combination with erlotinib (150 mg/day) was given in 3-week cycles. Figitumumab was administered as an IV infusion on study Days 1 and 2 in Cycle 1, and on Day 1 every 3 weeks (from Day 1) thereafter. Erlotinib was taken as 150 mg at least 1 hour before or 2 hours after the ingestion of food. Intent-to-treat population according to randomization was analyzed.
- Erlotinib (as Randomized): Erlotinib was taken as 150 mg daily at least 1 hour before or 2 hours after the ingestion of food. Intent-to-treat population according to randomization was analyzed.
- Total: Total of all reporting groups
Arm/Group | Figitumumab + Erlotinib (as Randomized) | Erlotinib (as Randomized) | Total
Number analyzed (Participants) | 293 | 290 | 583
Age, Customized [Number; unit: participants]
  <70 years | 226 | 222 | 448
  >=70 years | 67 | 68 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 65 | 130
  Male | 228 | 225 | 453

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The time from date of randomization to date of death due to any cause. For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline, assessed every cycle until disease progression and then every 4 weeks until death, up to 30.65 months
Population: Full (intent-to-treat) analysis set, which included all participants randomized regardless of treatment received.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Figitumumab + Erlotinib: Figitumumab (20 mg/kg) in combination with erlotinib (150 mg/day) was given in 3-week cycles. Figitumumab was administered as an IV infusion on study Days 1 and 2 in Cycle 1, and on Day 1 every 3 weeks (from Day 1) thereafter. Erlotinib was taken as 150 mg daily at least 1 hour before or 2 hours after the ingestion of food.
- Erlotinib: Erlotinib was taken as 150 mg daily at least 1 hour before or 2 hours after the ingestion of food.
Arm/Group | Figitumumab + Erlotinib | Erlotinib
Number analyzed (Participants) | 293 | 290
months | 5.7 [4.8 to 6.7] | 6.2 [5.8 to 7.2]
Statistical Analysis 1: Comparison: Figitumumab + Erlotinib vs Erlotinib; P-value was calculated using log-rank test stratified by gender (Male or Female), Eastern Cooperative Oncology Group (ECOG) performance status (less than or equal to [=<1] or 2), and region (United States/Canada, European Union, rest of world). The stratified Cox proportional hazards model was fitted to estimate the hazard ratio, using the same stratification variables as above; Test type: Superiority or Other; p = 0.35, Log Rank — One-sided significance level at alpha=0.024 was used. Two-sided p-value was reported; Nominal p-values were reported without adjustment for the interim analysis; Hazard Ratio (HR) = 1.091, 95% CI 2-sided [0.909 to 1.310]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from randomization to date of first documentation of progression or death due to any cause, whichever came first. Participants last known to be alive and progression-free, who had a baseline and at least 1 on-study disease assessment, were censored at last disease assessment verifying lack of progression. Progression was determined by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, as a 20% increase in the sum of the longest diameter of target lesions, or target lesions over nadir, unequivocal progression of non-target disease, or the appearance of new lesions.
Time Frame: Baseline, 6, 9, 12, 15, 18 weeks after randomization, thereafter assessed every 6 weeks until disease progression during treatment (or every 8 weeks until disease progression during off-treatment), up to 29.7 months
Population: Full (intent-to-treat) analysis set, which included all participants randomized regardless of treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Figitumumab + Erlotinib | Erlotinib
Number analyzed (Participants) | 293 | 290
months | 2.1 [1.9 to 2.6] | 2.6 [2.1 to 2.8]
Statistical Analysis 1: Comparison: Figitumumab + Erlotinib vs Erlotinib; P-value was calculated using log-rank test stratified by gender (Male or Female), ECOG performance status (less than or equal to [=<1] or 2), and region (United States/Canada, European Union, rest of world). The stratified Cox proportional hazards model was fitted to estimate the hazard ratio, using the same stratification variables as above; Test type: Superiority or Other; p = 0.426, Log Rank — One-sided significance level at alpha=0.001 was used. Two-sided p-value was reported; Hazard Ratio (HR) = 1.075, 95% CI 2-sided [0.898 to 1.287]

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response (OR) based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. CR are defined as complete disappearance of all lesions (target and/or non target). PR are those with at least 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: as for outcome 2
Population: Full (intent-to-treat) analysis set, which included all participants randomized regardless of treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Figitumumab + Erlotinib | Erlotinib
Number analyzed (Participants) | 293 | 290
percentage of participants | 5.5 [3.2 to 8.7] | 3.8 [1.9 to 6.7]
Statistical Analysis 1: Comparison: Figitumumab + Erlotinib vs Erlotinib; Test type: Superiority or Other; p = 0.338, Chi-squared; Difference in response rates = 1.668, 95% CI 2-sided [-1.7 to 5.1]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Figitumumab
Time Frame: Cycle 1 (Day 1 [predose], Day 2 [1 hour after end of infusion] ), Cycles 2, 4, 6 (predose), Cycle 5 (predose, 1 hour after end of infusion) for figi plus erlo group; Cycles 1, 2,4 (predose) for erlo, then figi group
Population: Due to futility, the study was terminated early; therefore pharmacokinetic data were not analyzed.
Groups:
- Figitumumab + Erlotinib, and Erlotinib Then Figitumumab: Participants who received figitumumab (20 mg/kg), whether figitumumab was given in combination with erlotinib (150 mg/day) from the beginning or figitumumab was given after disease progression with erlotinib (150 mg/day) alone. Figitumumab was administered as an IV infusion on study Days 1 and 2 in Cycle 1, and on Day 1 every 3 weeks (from Day 1) thereafter.
Arm/Group | Figitumumab + Erlotinib, and Erlotinib Then Figitumumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Figitumumab
Time Frame: as for outcome 4
Population: Due to futility, the study was terminated early; therefore pharmacokinetic data were not analyzed.
Arm/Group | Figitumumab + Erlotinib, and Erlotinib Then Figitumumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants Reporting Positive for Total Anti-drug Antibodies (ADA)
Description: ADAs are immunogenicity indicators to figitumumab. Participants reporting positive for ADAs are indicated by an endpoint titer of no less than 6.64.
Time Frame: Cycles 1, 2, 4 (predose), End of Treatment ([EOT] 21-28 days after last dose), about 150 days after last figi dose for figi plus erlo group; Cycles 1, 2, 4 (predose), EOT, about 150 days after last figi dose for erlo, then figi group
Population: Analysis population included all participants treated with figi. Data are combined for "figi+erlo" and "erlo then figi" because the objective was to report any participants with positive ADA after exposure to figi regardless of figi administration order, rather comparison of these 2 treatment groups. N=number of participants evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Figitumumab + Erlotinib, and Erlotinib Then Figitumumab
Number analyzed (Participants) | 360
percentage of participants | 0.28

7. Secondary Outcome: Counts of Circulating Tumor Cell (CTC) Expressing Positive Insulin-Like Growth Factor 1 Receptor (IGF-1R)
Time Frame: Baseline, Cycle 2 Day 1 (predose) and EOT (21-28 days after last dose)
Population: Due to futility, the study was terminated early; therefore biomarker results were not analyzed.
Arm/Group | Figitumumab + Erlotinib, and Erlotinib Then Figitumumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Euro Quality of Life (EQ-5D)- Health State Profile Utility at Cycles 2, 3, Then Every Other Cycle and EOT (21-28 Days After Last Dose)
Description: EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline (Cycle 1 Day 1 predose), Cycles 2, 3 (Day 1), every other cycle and EOT (21-28 days after last dose)
Population: Due to futility, the study was terminated early; therefore EQ-5D data were not analyzed.
Arm/Group | Figitumumab + Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30) at Cycles 2, 3, and Then Every Odd Cycle Starting With Cycle 5 and EOT (21-28 Days After Last Dose)
Description: EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions use 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline (Cycle 1 Day 1 predose), Cycles 2, 3 (Day 1), every odd cycle starting with Cycle 5 and EOT (21-28 days after last dose)
Population: This outcome measure was added in Protocol Amendment 3 (28 January 2010). However, data were not collected as the majority of the subjects had already been enrolled prior to this amendment and the study was terminated shortly thereafter (02 March 2010).
Arm/Group | Figitumumab + Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC), Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13) Score at Cycles 2, 3, and Then Every Odd Cycle Starting With Cycle 5, and EOT (21-28 Days After Last Dose)
Description: QLQ-LC13 consists of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprise 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain). Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: as for outcome 9
Population: as for outcome 9
Arm/Group | Figitumumab + Erlotinib | Erlotinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. All treated subjects were analyzed for AEs and SAEs.
Groups:
- Figitumumab + Erlotinib: Figitumumab (20 mg/kg) in combination with erlotinib (150 mg/day) was given in 3-week cycle. Figitumumab was administered as an IV infusion on study Days 1 and 2 in Cycle 1, and on Day 1 every three weeks (from Day 1) thereafter. Erlotinib was taken as 150 mg daily at least 1 hour before or 2 hours after the ingestion of food.
- Erlotinib, Then Figitumumab: Figitumumab (20 mg/kg) was given as a single agent after participants had disease progression on erlotinib alone. Figitumumab was given in 3-week cycles as IV infusion on study Days 1 and 2 in Cycle 1, and on Day 1 every 3 weeks (from Day 1) thereafter.
Arm/Group | Figitumumab + Erlotinib | Erlotinib | Erlotinib, Then Figitumumab
Serious Adverse Events (participants affected / at risk) | 204/289 | 153/290 | 63/83
Other Adverse Events (participants affected / at risk) | 265/289 | 265/290 | 79/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab + Erlotinib (N=289) | Erlotinib (N=290) | Erlotinib, Then Figitumumab (N=83)
Disease progression (General disorders) | 136 | 112 | 45
Dehydration (Metabolism and nutrition disorders) | 14 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 1
Pneumonia (Infections and infestations) | 9 | 12 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | 4 | 1
Asthenia (General disorders) | 5 | 1 | 0
Chest pain (General disorders) | 5 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Syncope (Nervous system disorders) | 5 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 2
Lower respiratory tract infection (Infections and infestations) | 4 | 0 | 1
Pyrexia (General disorders) | 4 | 5 | 1
Respiratory tract infection (Infections and infestations) | 4 | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 2
General physical health deterioration (General disorders) | 3 | 5 | 5
Pain (General disorders) | 3 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Death (General disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Band neutrophil count increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fungaemia (Infections and infestations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial strain (Investigations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Renal function test abnormal (Investigations) | 1 | 0 | 0
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pyothorax (Infections and infestations) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab + Erlotinib (N=289) | Erlotinib (N=290) | Erlotinib, Then Figitumumab (N=83)
Anaemia (Blood and lymphatic system disorders) | 28 | 26 | 11
Abdominal pain upper (Gastrointestinal disorders) | 8 | 8 | 5
Constipation (Gastrointestinal disorders) | 17 | 19 | 9
Diarrhoea (Gastrointestinal disorders) | 123 | 106 | 10
Dysphagia (Gastrointestinal disorders) | 14 | 11 | 6
Mouth ulceration (Gastrointestinal disorders) | 16 | 4 | 1
Nausea (Gastrointestinal disorders) | 54 | 36 | 8
Stomatitis (Gastrointestinal disorders) | 18 | 6 | 0
Vomiting (Gastrointestinal disorders) | 49 | 23 | 7
Asthenia (General disorders) | 79 | 46 | 25
Chest pain (General disorders) | 31 | 28 | 21
Fatigue (General disorders) | 65 | 53 | 16
Mucosal inflammation (General disorders) | 33 | 11 | 0
Oedema peripheral (General disorders) | 8 | 16 | 1
Pyrexia (General disorders) | 25 | 18 | 5
Paronychia (Infections and infestations) | 17 | 8 | 1
Weight decreased (Investigations) | 65 | 33 | 19
Decreased appetite (Metabolism and nutrition disorders) | 115 | 70 | 32
Dehydration (Metabolism and nutrition disorders) | 21 | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 37 | 13 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 11 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 25 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 9 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 5 | 1
Dizziness (Nervous system disorders) | 16 | 4 | 3
Headache (Nervous system disorders) | 13 | 14 | 9
Anxiety (Psychiatric disorders) | 7 | 7 | 6
Depression (Psychiatric disorders) | 10 | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 51 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 61 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 7 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 33 | 32 | 8
Acne (Skin and subcutaneous tissue disorders) | 9 | 17 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 22 | 14 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 30 | 24 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 31 | 3
Rash (Skin and subcutaneous tissue disorders) | 140 | 152 | 33
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 4 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0
Atrial flutter (Cardiac disorders) | 0 | 2 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 4 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 4 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 2 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 2 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Blindness (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 10 | 14 | 2
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 5 | 1
Eye inflammation (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 2 | 0 | 0
Eye pain (Eye disorders) | 1 | 2 | 1
Eye pruritus (Eye disorders) | 4 | 3 | 1
Eye swelling (Eye disorders) | 0 | 2 | 0
Eyelid oedema (Eye disorders) | 2 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 3 | 0 | 0
Lacrimation increased (Eye disorders) | 5 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0
Ocular toxicity (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 3 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 9 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 1
Aerophagia (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 3 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 8 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Gingival disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 2 | 2
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 2 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 1
Oral pain (Gastrointestinal disorders) | 4 | 2 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 1 | 0
Retching (Gastrointestinal disorders) | 2 | 0 | 0
Salivary gland disorder (Gastrointestinal disorders) | 1 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Tooth socket haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Axillary pain (General disorders) | 1 | 1 | 0
Chest discomfort (General disorders) | 4 | 2 | 0
Chills (General disorders) | 4 | 3 | 1
Disease progression (General disorders) | 6 | 4 | 3
Early satiety (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 2 | 2 | 0
Facial pain (General disorders) | 0 | 1 | 0
Feeling cold (General disorders) | 2 | 1 | 0
Gait disturbance (General disorders) | 2 | 0 | 0
General physical health deterioration (General disorders) | 4 | 1 | 0
Hyperthermia (General disorders) | 1 | 3 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 0 | 1 | 1
Localised oedema (General disorders) | 0 | 3 | 0
Malaise (General disorders) | 2 | 1 | 1
Medical device pain (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 2 | 1 | 0
Pain (General disorders) | 5 | 7 | 3
Performance status decreased (General disorders) | 2 | 0 | 1
Ulcer (General disorders) | 1 | 0 | 0
Xerosis (General disorders) | 1 | 5 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 4 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 5 | 0 | 0
Acne pustular (Infections and infestations) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 7 | 3
Candidiasis (Infections and infestations) | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 3 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 1 | 1
Eye infection bacterial (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 2 | 0
Fungal infection (Infections and infestations) | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 3 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 3 | 1
Lung infection (Infections and infestations) | 5 | 3 | 2
Mediastinitis (Infections and infestations) | 0 | 0 | 1
Nail bed infection (Infections and infestations) | 1 | 0 | 0
Nail infection (Infections and infestations) | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Omphalitis (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 4 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 6 | 3 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pyothorax (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 4 | 2 | 1
Respiratory moniliasis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 3 | 2
Rhinitis (Infections and infestations) | 3 | 3 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 2
Skin candida (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 2 | 0 | 0
Sputum purulent (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 1
Urethritis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 8 | 6 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 1 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 2 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 7 | 10 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 10 | 1
Blood alkaline phosphatase increased (Investigations) | 6 | 7 | 0
Blood bilirubin increased (Investigations) | 2 | 3 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood creatine increased (Investigations) | 4 | 0 | 0
Blood creatinine increased (Investigations) | 12 | 3 | 3
Blood glucose increased (Investigations) | 3 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 4 | 0
Blood magnesium decreased (Investigations) | 3 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 3 | 3 | 1
Blood urea nitrogen/creatinine ratio increased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 4 | 0 | 2
Body temperature increased (Investigations) | 1 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 4 | 2 | 4
Breath sounds abnormal (Investigations) | 0 | 1 | 1
Clostridium test positive (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 13 | 6 | 3
General physical condition abnormal (Investigations) | 3 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 2
Liver function test abnormal (Investigations) | 2 | 0 | 0
Nutritional condition abnormal (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Protein urine (Investigations) | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 1
Prothrombin time shortened (Investigations) | 0 | 1 | 0
Renal function test abnormal (Investigations) | 1 | 0 | 0
Respiratory rate decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 0 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 6 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 4 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 7 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 2
Ageusia (Nervous system disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 1
Aphonia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 2 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 4 | 0 | 3
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 12 | 5 | 4
Dyskinesia (Nervous system disorders) | 2 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 2 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 3 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 1
Monoparesis (Nervous system disorders) | 0 | 1 | 1
Movement disorder (Nervous system disorders) | 0 | 1 | 0
Myotonia (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 4 | 0
Paraesthesia (Nervous system disorders) | 5 | 8 | 2
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 4 | 2 | 1
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 2 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Tremor (Nervous system disorders) | 1 | 0 | 2
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 3 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 1
Affective disorder (Psychiatric disorders) | 0 | 2 | 2
Agitation (Psychiatric disorders) | 1 | 1 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 10 | 3 | 2
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Dysthymic disorder (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 12 | 8 | 3
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 3 | 3
Dysuria (Renal and urinary disorders) | 5 | 1 | 2
Haematuria (Renal and urinary disorders) | 2 | 2 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 8 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 6 | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2 | 2
Balanitis (Reproductive system and breast disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 3
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 6 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 3 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 8 | 5 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 10 | 6 | 1
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 3 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 6 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 11 | 9 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Surgical and medical procedures) | 0 | 1 | 1
Hot flush (Vascular disorders) | 3 | 0 | 0
Hypertension (Vascular disorders) | 10 | 3 | 2
Hypotension (Vascular disorders) | 13 | 7 | 2
Orthostatic hypotension (Vascular disorders) | 4 | 0 | 0
Phlebitis (Vascular disorders) | 2 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.